CLINICAL TRIAL: NCT06698471
Title: Relief From Stress Via Social Protection in Senegal (RESTORE): Study Protocol for a Pilot Feasibility Cluster-randomized Control Trial of Self-Help Plus (SH+) in Senegal.
Brief Title: Relief From Stress Via Social Protection in Senegal
Acronym: RESTORE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: World Bank (Other); Centre de Recherche Pour le Développement Economique et Social (CRDES) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB#2575
Record Dates: First submitted 2024-10-22; First posted 2024-11-21 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-03

CONDITIONS: Distress, Psychological; Depression - Major Depressive Disorder; Generalized Anxiety Disorder (GAD)
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcome assessors are masked to study arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as usual (Active Comparator): Treatment as usual from Health System in Senegal
  Interventions: Other: Referral to Health System
- Relief from Stress via Social Protection in Senegal (Experimental): Training community workers in Self Help Plus intervention
  Interventions: Other: Community worker training

INTERVENTIONS:
Other: Community worker training — Training community workers in Self Help Plus intervention, a 5 session self-help intervention based on Acceptance and Commitment Therapy
  Arms: Relief from Stress via Social Protection in Senegal
Other: Referral to Health System — Referral to Health System of Senegal
  Arms: Treatment as usual

SUMMARY:
Despite the growing prevalence of mental health disorders in low- and middle-income countries, significant barriers to seeking and accessing mental health services persist. Within lower income populations, the prevalence of mental health disorders and barriers to addressing them are worsened by poverty. Self-Help Plus is a group-based stress management program delivered using a task-sharing model and designed to circumvent barriers to addressing mental health concerns. Cultural adaptations of Self-Help Plus have been implemented in several countries and are considered cost-effective. However, to date, Self-Help Plus has not been adapted for Senegalese populations. The study detailed in this manuscript aims to assess the feasibility and acceptability of Self-Help Plus in lower income populations in Senegal.

The study is a pilot feasibility cluster-randomized control trial of Self-Help Plus in four Senegalese communities. Clusters of social protection program beneficiaries will be randomly selected to receive five sessions of Self-Help Plus. The intervention will be delivered in groups of up to 30 beneficiaries and co-facilitated by two community workers. A combination of quantitative and qualitative research methods will be used to assess the feasibility and acceptability of both the Self-Help Plus intervention and randomized control trial procedures. The study sample will include social protection program beneficiaries in the treatment and control groups, Self-Help Plus facilitators, project staff supporting the training of facilitators, and the intervention supervisor.

The findings of this study will be used to inform the potential integration of Self-Help Plus and/or similar mental health interventions into the national social protection program in Senegal.

DETAILED DESCRIPTION:
The primary objective of the pilot feasibility cluster-randomized controlled trial is to assess the feasibility and acceptability of both the Self-Help Plus intervention and trial procedures through the collection of quantitative and qualitative data. The study will include two trial arms: (1) a control treatment-as-usual arm and (2) an intervention arm that will receive the adapted Self Help Plus intervention. The findings of the research detailed in this protocol may be used to inform the design of a potential larger randomized control trial powered to assess the effectiveness of Self-Help Plus in Senegalese populations. Additional secondary objectives of the pilot feasibility study are listed below.

1. Assess feasibility of cluster randomization procedure to limit biases and risk of contamination;
2. Determine recruitment and retention rates for Self-Help Plus sessions;
3. Evaluate the feasibility and acceptability of intervention delivery by Self-Help Plus trained non-specialists;
4. Assess the safety of an abbreviated training curriculum (during training, intervention delivery, and supervision);
5. Assess feasibility and acceptability of outcome measures;
6. Assess ethics and safety of trial procedures using the adverse event protocol;

ELIGIBILITY:
Inclusion Criteria:

* Community Worker facilitators of the intervention:
* Patients: Enrolled in the World Bank Social Protection Programme

Exclusion Criteria:

* Community Worker facilitators of the intervention
* Patients: Persons with a severe mental disorder or suicidality

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 748 (Actual)
Dates: Start 2025-02-24 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Engagement | From enrollment to the end of treatment at 5 weeks
  Of those who were offered the intervention, at least 25% attended one or more sessions.
Retention | From enrollment to the end of treatment at 5 weeks
  At least 50% of the ever-attended beneficiaries attended at least any 4 intervention sessions
Fidelity | From enrollment to the end of treatment at 5 weeks
  Fidelity to intervention elements at the level of 75% or greater according to the mean fidelity checklist for intervention elements across all sessions. Number of feasibility domains: n=15; higher is better, scored on 0-100%

SECONDARY OUTCOMES:
General Health Questionnaire-12 | Prior to initiation of treatment
  Brief psychological well-being scale. Score range: 0-36; Higher score indicates worse psychological well-being
General Health Questionnaire-12 | 2 months following initiation of treatment
  Brief psychological well-being scale. Score range: 0-36; Higher score indicates worse psychological well-being
General Health Questionnaire-12 | 5 months following initiation of treatment
  Brief psychological well-being scale. Score range: 0-36; Higher score indicates worse psychological well-being
Patient Health Questionnaire-9 | Prior to initiation of treatment
  Brief depression screening instrument. Score range: 0-27; Higher score indicates worse depressive symptoms
Patient Health Questionnaire-9 | 2 months following initiation of treatment
  Brief depression screening instrument. Score range: 0-27; Higher score indicates worse depressive symptoms
Patient Health Questionnaire-9 | 5 months following initiation of treatment
  Brief depression screening instrument. Score range: 0-27; Higher score indicates worse depressive symptoms
Generalized Anxiety Disorder-7 | Prior to initiation of treatment
  Brief anxiety screening instrument. Score range: 0-21; Higher score indicates worse anxiety symptoms
Generalized Anxiety Disorder-7 | 2 months following initiation of treatment
  Brief anxiety screening instrument. Score range: 0-21; Higher score indicates worse anxiety symptoms
Generalized Anxiety Disorder-7 | 5 months following initiation of treatment
  Brief anxiety screening instrument. Score range: 0-21; Higher score indicates worse anxiety symptoms
Brief Resilience Scale | Prior to initiation of treatment
  Brief resilience measure. Score range: 0-30; Higher score indicates better resilience
Brief Resilience Scale | 2 months following initiation of treatment
  Brief resilience measure. Score range: 0-30; Higher score indicates better resilience
Brief Resilience Scale | 5 months following initiation of treatment
  Brief resilience measure. Score range: 0-30; Higher score indicates better resilience
Acceptance and Action Questionnaire | Prior to initiation of treatment
  Brief scale of psychological flexibility. Score range: 0-35; Higher score indicates worse psychological flexibility
Acceptance and Action Questionnaire | 2 months following initiation of treatment
  Brief scale of psychological flexibility. Score range: 0-35; Higher score indicates worse psychological flexibility
Acceptance and Action Questionnaire | 5 months following initiation of treatment
  Brief scale of psychological flexibility. Score range: 0-35; Higher score indicates worse psychological flexibility
Self Efficacy | Prior to initiation of treatment
  Brief scale of self efficacy. Score range: 0-24; Higher score indicates better self efficacy
Self Efficacy | 2 months following initiation of treatment
  Brief scale of self efficacy. Score range: 0-24; Higher score indicates better self efficacy
Self Efficacy | 5 months following initiation of treatment
  Brief scale of self efficacy. Score range: 0-24; Higher score indicates better self efficacy
Locus of control questionnaire | Prior to initiation of treatment
  Brief scale measuring locus of control. Score range: 0-20; Higher score indicates better locus of control
Locus of control questionnaire | 2 months following initiation of treatment
  Brief scale measuring locus of control. Score range: 0-20; Higher score indicates better locus of control
Locus of control questionnaire | 5 months following initiation of treatment
  Brief scale measuring locus of control. Score range: 0-20; Higher score indicates better locus of control

OTHER OUTCOMES:
Culture-specific measure of distress - Thinking too much | Prior to initiation of treatment
  Exploratory 1-item culture-specific measure of distress; Score range: 0-5; Higher score indicates worse psychological well-being
Culture-specific measure of distress - Thinking too much | 2 months following initiation of treatment
  Exploratory 1-item culture-specific measure of distress; Score range: 0-5; Higher score indicates worse psychological well-being
Culture-specific measure of distress - Thinking too much | 5 months following initiation of treatment
  Exploratory 1-item culture-specific measure of distress; Score range: 0-5; Higher score indicates worse psychological well-being
Culture-specific measure of distress - Feelings that hurt the heart | Prior to initiation of treatment
  Exploratory 1-item culture-specific measure of distress; Score range: 0-5; Higher score indicates worse psychological well-being
Culture-specific measure of distress - Feelings that hurt the heart | 2 months following initiation of treatment
  Exploratory 1-item culture-specific measure of distress; Score range: 0-5; Higher score indicates worse psychological well-being
Culture-specific measure of distress - Feelings that hurt the heart | 5 months following initiation of treatment
  Exploratory 1-item culture-specific measure of distress; Score range: 0-5; Higher score indicates worse psychological well-being
Culture-specific measure of well being - Heart has felt calm | Prior to initiation of treatment
  Exploratory 1-item culture-specific measure of well being; Score range: 0-3; Higher score indicates better well being
Culture-specific measure of well being - Heart has felt calm | 2 months following initiation of treatment
  Exploratory 1-item culture-specific measure of well being; Score range: 0-3; Higher score indicates better well being
Culture-specific measure of well being - Heart has felt calm | 5 months following initiation of treatment
  Exploratory 1-item culture-specific measure of well being; Score range: 0-3; Higher score indicates better well being

CONTACTS AND LOCATIONS:
Overall Officials: Syed S Wahid, Doctor of Public Health, Principal Investigator — Georgetown University; Anne Hilger, PhD, Principal Investigator — World Bank
Locations (1):
- Centre de Recherche Pour le Développement Economique et Social (CRDES), Dakar, Senegal

IPD SHARING:
Plan to Share IPD: Undecided